CLINICAL TRIAL: NCT02903550
Title: Usefulness of Non EPI-DWI-MRI / CT 3D Static Co-registration Prior to Surgery of Cholesteatomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-27
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Cholesteatoma
MeSH Terms: conditions — Cholesteatoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cholesteatoma is a destructive and expanding pathologic condition consisting of keratin pearl arising from a squamous epithelium in the middle ear and/or mastoid process. Evolution consists in a destruction of the ossicles as well as their possible spread through the base of the skull into the brain. Surgical treatment is required to prevent infectious or functional complications. A recurrence after surgery occurs in approximately 10% of patients and rarely affects initial site. Surgical treatment is the only care option for recurrent cholesteatoma. Various locations such as surgical approach cavity, mastoid, hypotympanum are seen. Temporal bone CT is performed prior to surgery for added information on bone erosions especially of ossicules, tegmen tympani, facial nerve canal of internal ear. Due high anatomical resolution and complex anatomy, temporal bone CT is usually displayed with Magnetic Resonance Imaging (MRI) in operating room to help surgical guidance .

Imaging especially using MRI is the cornerstone for diagnosis in asymptomatic patients. Since 2006, non echo planar imaging (EPI) Diffusion weighted imaging (DWI) Magnetic resonance imaging (MRI) (sequences has shown high accuracy to depict recurrent cholesteatoma. If EPI sequences had a high rate of diffeomorphic atefacts whereas non EPI sequences using either HAlf-Fourier acquisition Single-shot Turbo spin-Echo (HASTE) or Fast-spin-echo demonstrates less magnetic susceptibility artifacts. Multimodality fusion between NonEPI-DWI-MRI and computerized tomography (CT) is a rational promising tool to rise the performance for cholesteatomas delineation. The performances of NonEPI-DWI-MRI in assessing lesion spread and volume are still unknown and needs further investigations. The aim of the study is to assess the DWI-MRI/CT fusion feasibility, reproducibility and the accuracy prior to surgery propectively compared to surgical findings.

ELIGIBILITY:
Inclusion Criteria:

- Adult woman or man who had surgery and suspicion of cholesteatoma recurrence

Exclusion Criteria:

* Chronic renal failure
* Contraindications to MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who had surgery and suspicion of recurrence of cholesteatoma for whom it is prescribed:
  * MRI with diffusion through systematic monitoring after treatment of acquired cholesteatoma of the middle ear: between 12 and 18 months and 4 years
  * If positive MRI scanner producing a rock without injection in the preoperative assessment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Determination of the lesion on the scanner with the help of MRI, but without having merged both methods | UP to 18 months
Measure of the lesion volume in mm3 | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de La Timone - Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided